CLINICAL TRIAL: NCT00795743
Title: The Effect of Central Venous Catheters on Systemic Coagulation
Brief Title: Coagulation Changes in Trauma Patients
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Kenneth Proctor, Professor, University of Miami
Other Study IDs: 20070692
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Deep Vein Thrombosis
Keywords: Central Venous Catheterization; coagulopathy; thromboelastography
MeSH Terms: conditions — Venous Thrombosis; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis to be tested: placement of a central venous catheter will induce a systemic hypercoagulable state. To determine this, the investigators will measure thromboelastography (TEG), PT(prothrombin time), PTT (partial thromboplastin time), Prothrombin Fragment 1.2, Factor VIII, and VonWillebrand's Factor. In addition, duplex ultrasound will be performed to correlate the laboratory coagulation values with functional changes (i.e. deep venous thrombosis).

DETAILED DESCRIPTION:
We will enroll all patients who will be getting a Central Venous Catheter (CVC) placed either in the PICC Insertion Room or in a surgical intensive care unit who are undergoing emergent central venous catheter placement for a medically indicated reason. All patients who have not had a previous central line or will be getting their catheter exchanged over guide wire are eligible.

At Baseline:

We intend to evaluate the patient for a Deep Vein Thrombosis by conducting a duplex ultrasound of the lower extremities prior to line insertion. We will also collect one sample of blood at baseline within 3 hours of insertion.

During CVC Insertion:

One sample of blood will be collected during CVC insertion.

Follow Up:

The last blood sample will be collected soon after CVC insertion (approximately 3hrs). Blood samples will only be drawn when we are available to collect them. Thus, this is defined as a "sample of convenience". We will also conduct another duplex ultrasound of the extremities after CVC insertion for evaluation of DVT.

Data will be collected on the duplex ultrasound result, the type of central line and the exact insertion site. Should a DVT be found, the attending physician will be made aware according to clinical protocol.

Normally, at the moment of central venous puncture, 5cc of blood is aspirated and wasted to confirm correct placement of the needle tip before placement of the guidewire. For the intended study, instead of wasting that blood, we will save 500 microliters of it for coagulation analysis. Immediately after the catheter is inserted over the guidewire, a chest x-ray is obtained to verify position of the catheter. At this point, each port of the central venous catheter is aspirated and wasted before infusion through the central venous catheter. For the purpose of this study, we will save 500 microliters of that wasted blood for coagulation analysis. To clarify, the second 500 microliters will be drawn through the newly placed central venous catheter ports and saved (instead of being drawn and wasted). Drawing back on each port before infusing is standard practice. This second sample will contain a small amount of saline, but, based on a few trials in the animal lab, this saline is unlikely to effect the coagulation analysis.

In summary, we intend to visit the patient 3 times over approximately a 4 hour period for the purpose of collecting blood that would normally otherwise be wasted (a total of 1500 microliters). This will be done only on patients who are undergoing the procedure for for a medically indicated reason and medical care will not be changed, affected, or otherwise altered based on involvement in this study. Our purpose is simply to collect 3 samples of blood during emergent central venous catheter placement that would otherwise be wasted into the biohazard container.

We will use this blood to assay prothrombin time, partial thromboplastin time, thromboelastography, Prothrombin Fragment 1.2, Factor VIII, and VonWillebrand's Factor.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing placement of a central venous catheter.

Exclusion Criteria:

* Age under 18 or known coagulation disorder (inherited or pharmacologic).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PAtients requiring placement of a central venous catheter.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Coagulopathy | 3 hours surrounding placement of catheter

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G Proctor, PhD, Principal Investigator — University of Miami
Locations (1):
- Ryder Trauma Center, Miami, Florida, United States

REFERENCES:
- [Background] King DR, Cohn SM, Feinstein AJ, Proctor KG. Systemic coagulation changes caused by pulmonary artery catheters: laboratory findings and clinical correlation. J Trauma. 2005 Oct;59(4):853-7; discussion 857-9. doi: 10.1097/01.ta.0000187656.26849.39. PMID 16374273